CLINICAL TRIAL: NCT02614599
Title: Neurocognitive and Neurobiological Improvement in ADHD Children by Modification of Dietary Protein
Brief Title: Neurocognitive and Neurobiological Improvement in ADHD Children With High Protein Diet
Acronym: BrainProtein
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Spanish Foundation for Neurometrics Development (Other)
Collaborators: PronoKal Foundation (Other); Child Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BrainProteins
Record Dates: First submitted 2013-04-22; First posted 2015-11-25 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2015-11

CONDITIONS: ADD; ADHD
Keywords: ADD; ADHD; Proteins; Dietary; Nutrition; QEEG; ERP; ICA
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BP22042013 (Experimental): This group of patients receive 2.000 kilocalories diet(60 g. carbohydrates, 144 gr of fat and 107 gr of proteins), including 2 protein shakes.
  Interventions: Drug: BP22042013
- Low carbohydrate Diet (Experimental): the second group of patients receive diet of 2.000 Kilo calories without rapidly absorbed carbohydrates and without proteins supplements
  Interventions: Dietary Supplement: Low carbohydrate diet

INTERVENTIONS:
Drug: BP22042013 — This group of patients receive 2.000 kilo-calories diet (60 g. carbohydrates, 144 gr of fat and 107 gr of proteins), including 2 protein shakes.
  Other Names: Brain Proteins Supplements
  Arms: BP22042013
Dietary Supplement: Low carbohydrate diet — the second group of patients receive diet of 2.000 Kilo-calories without rapidly absorbed carbohydrates and without proteins supplements
  Other Names: 2000 Kilo-calories without Fast Absorbing Carbohydrate
  Arms: Low carbohydrate Diet

SUMMARY:
Multicenter, Prospective, randomized, comparative and controlled study about the beneficial effects in behavior and brain connectivity of different dietary patterns in 100 children with ADHD between 7 and 12 years, followed up for 3 months of nutritional therapy.

DETAILED DESCRIPTION:
We collect electroencephalogram (EEG), event related potentials (ERP) data, and behavior parameters in ADD/ADHD children that not take stimulants or other drugs during study. They would only follow some nutritional recommendations based on increasing the amount of dietary protein and fast carbohydrates decrease. The duration of the study will be 6 months, 3 months for recruitment and 3 months for dietary treatment.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosed 12 months before
* no take medication
* BMI above the 25th percentile
* Wiesel score between 80 and 100 (about 120)
* Patients who agree to participate and whose guardians signed the informed consent form

Exclusion Criteria:

* eating disorders
* psychosis, bipolar disorder or depression
* kidney or liver failure
* diabetes
* diuretic or cortisone treatment
* haematological problems
* suprarenal diseases
* cancer
* Brain injury
* Cardiovascular or arrhythmia problems

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes Related Potential Recording after 3 months of dietary approach | 3 months
  Evaluate changes in reaction time, omission and comission errors, latencies and amplitudes in brainwaves during visual continuous performance task from 19 channels EEG recordings, before begin nutritional measures and after 3 months of dietary approach.

SECONDARY OUTCOMES:
Quantitative Electroencephalogram | 3 months
  Analysis frequencies and amplitudes of brainwaves and spectral independent components before and after 3 months of nutritional intervention
Behavior | 3 months
  Evaluate Behavior with clinical scales (AMEN questionnaire) at the beginning and after 3 months of nutritional approach.

OTHER OUTCOMES:
Change in Weight | 3 months
  Change from Baseline in Weight after 3 months of nutritional intervention
Change in body mass index | 3 months
  Change in body mass index after 3 months of nutritional intervention.
Change in body composition | 3 months
  Change in body composition using bioelectrical impedance after 3 months of nutritional intervention.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From April to December 2013
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability of Brain Proteins Supplements

REFERENCES:
- See also: Brainmech Foundation — http://www.brainmech.org
- See also: Neurometrics — http://www.qeeg.es
- See also: Children Health Foundation — http://www.fundacionsaludinfantil.org